CLINICAL TRIAL: NCT03707327
Title: Effect of Two Methods for the Application of Cryotherapy in Pain and Surface Temperature of the Skin in Women With Previous Pain in the Knee
Brief Title: Effect of Two Methods for the Application of Cryotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Knee Cryotherapy Technique
Record Dates: First submitted 2018-07-23; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-07

CONDITIONS: Pain
Keywords: pain; knee; cryotherapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game Ready group (Experimental): the participants performed cryotherapy by compression with Game Ready
  Interventions: Other: Game Ready
- Ice pack (Experimental): the participants performed cryotherapy for ice pack
  Interventions: Other: Ice pack

INTERVENTIONS:
Other: Game Ready — the participants remained for 20 minutes with intermittent compression therapy + cryotherapy
  Arms: Game Ready group
Other: Ice pack — the participants remained for 20 minutes with cryotherapy with ice pack
  Arms: Ice pack

SUMMARY:
Introduction: Little is known about the effects of different cryotherapy techniques for pain and skin surface temperature in patients with anterior knee pain. Objective: To analyze the best technique of cryotherapy intervention to reduce the superficial temperature of the skin and pain of women with anterior pain in the knee. Methodology: The sample will be composed of 12 participants, of the female gender, aged between 18 and 25 years old and complaint of anterior pain in the knee, distributed in cryotherapy groups by ice pack (CPG) (n = 6) and cryotherapy + compression group byGame Ready (CCGR) (n = 6). All will complete the consent form, the sample characterization form, the Visual Analog Pain Scale (EVA) and the Patellofemoral Disorders Scale (AKPS). They will then have the basal temperature of the anterior knee region recorded by thermographic camera and perform five repetitions of the sit and stand test in 30 seconds. The EVA will again respond and the temperature of the anterior knee region will be collected after the test. Subsequently, CPG or CCGR (randomly) will be applied to the anterior region of the knee for 20 minutes. Immediately after the application of cryotherapy, EVA will be applied and will have the skin surface temperature recorded immediately after, and at 10, 20, 30 and 60 minutes. Expected results: It is expected to establish if there is difference in pain, surface temperature and skin reheating of women submitted to cryotherapy by ice pack and Game Ready.

DETAILED DESCRIPTION:
After the contact, explanation of the study procedures and acceptance of the participants, the data collection will be started and performed in the teaching laboratory of the Physiotherapy course of the State University of Londrina.

Initially, the demographic data of the sample (age, height, weight, limb and time of pain) and signature of the consent term will be collected.

After this step, the participants should point to the Visual Analogue Scale (EVA) and the Patellofemoral Disorders Scale (AKPS). Before performing the cryotherapy technique, the basal skin temperature in the anterior region of the knee will be recorded by means of a thermographic camera, and the participants will be submitted to five sets of the sit and stand test in 30 ', with rest of one minute between them. They will then re-signal the EVA and the skin temperature will be retained by the camera. Finally, they will undergo the application of cryotherapy according to the category which has been "randomized".

The two different intervention techniques will be:

* Ice pack group (CPG): where the participant will have a plastic bag containing 500 grams of crushed ice over the anterior region of the knee, and lie flat with the lower limb extended and supported on the ground for 20 minutes;
* Group Cryotherapy + Compression by Game Ready® (CCGR): where the participant will have the knee joint wrapped and compressed by the equipment where temperature, compression and time will be controlled, maximum compression, for 20 minutes by the equipment itself; lie in the same manner as for the other intervention.

Immediately thereafter, the EVA will be applied and the skin surface temperature recorded in the knee region, as well as 10, 20, 30 and 60 minutes thereafter.

ELIGIBILITY:
Inclusion Criteria:

* women
* anterior knee pain

Exclusion Criteria:

* muscle or joint injuries in the last month
* vascular problems
* allergy to cold
* lower limb surgery in the last 6 months
* viral conditions (such as colds or flu)

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-10-20 (Estimated); Primary Completion 2019-04-20 (Estimated); Study Completion 2019-09-20 (Estimated)

PRIMARY OUTCOMES:
Pain | preheating
  measurement pain by analogue visual scale (Score zero to ten, when zero is painless and 10 is maximum pain)
Pain | pre-intervention
  measurement pain by analogue visual scale (Score zero to ten, when zero is painless and 10 is maximum pain)
Pain | immediately post-intervention
  measurement pain by analogue visual scale (Score zero to ten, when zero is painless and 10 is maximum pain)
Pain | up to 60 minutes
  measurement pain by analogue visual scale (Score zero to ten, when zero is painless and 10 is maximum pain)

SECONDARY OUTCOMES:
Temperture | preheating
  through thermographic camera
Temperture | pre-intervention
  through thermographic camera
Temperture | immediately post-intervention
  through thermographic camera
Temperture | after 10 minutes
  through thermographic camera
Temperture | after 20 minutes
  through thermographic camera
Temperture | after 30 minutes
  through thermographic camera
Temperature | after 60 minutes
  through thermographic camera

CONTACTS AND LOCATIONS:
Overall Officials: Christiane G Macedo, PhD, Principal Investigator — State University of Londrina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey DM, Erith SJ, Griffin PJ, Dowson A, Brewer DS, Gant N, Williams C. Influence of cold-water immersion on indices of muscle damage following prolonged intermittent shuttle running. J Sports Sci. 2007 Sep;25(11):1163-70. doi: 10.1080/02640410600982659. PMID 17654228
- [Background] Bleakley C, McDonough S, Gardner E, Baxter GD, Hopkins JT, Davison GW. Cold-water immersion (cryotherapy) for preventing and treating muscle soreness after exercise. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD008262. doi: 10.1002/14651858.CD008262.pub2. PMID 22336838